CLINICAL TRIAL: NCT00569361
Title: Nasal Epithelium Gene Expression Profiling in Child Respiratory Allergic
Brief Title: Nasal Epithelium Gene Expression Profiling in Child Respiratory Allergic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: ADPHUN, FRM (Unknown)
Responsible Party: Département de la Recherche Clinique et de l'Innovation, CHU de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIR 2005
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis to dust mite; allergic rhinitis associated with bronchial hyperreactivity; allergic rhinitis associated with asthma
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Collection of nasal epithelial cells by brushing
  Interventions: Procedure: Collection of nasal epithelial cells

INTERVENTIONS:
Procedure: Collection of nasal epithelial cells — Collection of nasal epithelial cells by brushing

SUMMARY:
Using a human pangenomic microarray, the researchers established expression profiles of nasal epithelial cells, collected by brushing of patients belonging to one of four distinct groups:

1. allergic rhinitis to dust mite (AR) isolated (n=12),
2. AR associated with bronchial hyperreactivity (n=12),
3. AR associated with asthma (n=14),
4. control (n=14).

DETAILED DESCRIPTION:
Context: Asthma is the most frequent chronic disease in childhood. Allergic rhinitis has been described as a risk factor to develop asthma. The objective of the study was to evaluate the contribution of the respiratory epithelium to development of allergic rhinitis and asthma and to identify the molecular mechanisms driving rhinitis toward asthma.

Methods: Using a human pangenomic microarray, we established expression profiles of nasal epithelial cells, collected by brushing of patients belonging to one of four distinct children 2 to 18 years of age groups:

1. allergic rhinitis to dust mite (AR) isolated (n=12),
2. AR associated with bronchial hyperreactivity (n=12),
3. AR associated with asthma (n=14),
4. control (n=14).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients between 6 and 17 years old
* Patients with allergic rhinitis

Witness:

* Patients between 6 and 17 years old
* Patients without allergic rhinitis and asthma

Exclusion Criteria:

* Rhino-bronchitis infection dated from less than 15 days
* Patients younger than 6 or older than 17 years

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2004-11; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Transcriptome analysis: genes statistically modulated between groups, predictive biomarkers allowing correct classification of groups | At the sample time

SECONDARY OUTCOMES:
Validation with other techniques: Q-PCR | At the sample time

CONTACTS AND LOCATIONS:
Overall Officials: Marc Albertini, Professor, Principal Investigator — Department of Pediatrics of Nice University Hospital
Locations (1):
- Department of Pediatrics, Nice University Hospital, Nice, France

REFERENCES:
- [Derived] Giovannini-Chami L, Marcet B, Moreilhon C, Chevalier B, Illie MI, Lebrigand K, Robbe-Sermesant K, Bourrier T, Michiels JF, Mari B, Crenesse D, Hofman P, de Blic J, Castillo L, Albertini M, Barbry P. Distinct epithelial gene expression phenotypes in childhood respiratory allergy. Eur Respir J. 2012 May;39(5):1197-205. doi: 10.1183/09031936.00070511. Epub 2011 Oct 17. PMID 22005912